CLINICAL TRIAL: NCT00395681
Title: Population Pharmacokinetics and Pharmacodynamics of Propofol in the Morbidly Obese Patient
Brief Title: Population PK/PD of Propofol in the Morbidly Obese Patient
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Responsible Party: S. van Kralingen, St. Antonius Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13980
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2006-11

CONDITIONS: Morbid Obesity
Keywords: Obesity; Propofol; Morbidly obese; BMI
MeSH Terms: conditions — Obesity, Morbid; Obesity | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- propofol (Active Comparator): propofol 200 mg versus 350 mg
  Interventions: Drug: Diprivan
- Propofol (Active Comparator): Propofol 350 mg versus 200 mg
  Interventions: Drug: Diprivan

INTERVENTIONS:
Drug: Diprivan — Propofol 200 mg versus 350 mg

SUMMARY:
Rationale: The extreme increase of obesity in the last years had led to this study. There is no consensus about how to anaesthetise morbidly obese patients. The amounts of narcotics given vary widely and rather depend on the anaesthetist than on the pharmacokinetics and dynamics in the morbidly obese patient. Reason for this is that it is not clear in what extend the pharmacokinetics and dynamics are affected in the morbidly obese patient.

Objective: The study is performed in order to develop a population pharmacokinetic and pharmacodynamic model of Propofol when used for induction and maintenance of anaesthesia in the morbidly obese patient (BMI > 40). A covariate analysis will be performed in order to account for variability in pharmacokinetic and/or pharmacodynamic parameters. This model will take into account patient and procedure bound covariates. The results will be used to develop individualised dosing schemes of Propofol when used for induction and maintenance of anaesthesia in morbidly obese patients.

Study design: A randomised, therapeutic and non-invasive study.

Study population: Morbidly obese patients with a Body Mass Index > 40 undergoing laparoscopic banding or gastric bypass surgery, 18-60 year old.

Intervention (if applicable): Patients will be randomised into two groups, one group will be given 200 milligrams of Propofol and the other group will be given 350 milligrams of Propofol. During the induction of anaesthesia with Propofol over 60 seconds, the patient is asked to count in order to measure time to induction of anaesthesia. During and following anaesthesia a maximum of 50 ml of blood will be taken from an indwelling arterial line. Depth of sedation will be measured using non-invasive Bispectral Index (target 40-60) and other standard measures (heart frequency and blood pressure).

Main study parameters/endpoints: Primary endpoints: pharmacokinetic parameters; clearance, intercompartmental clearance, volume of central compartment and volume of peripheral compartment.

Secondary endpoints: pharmacodynamic parameters; time to induction of anaesthesia (stop counting, eyelash reflex, quality of anaesthesia, corresponding dose required for induction of anaesthesia for both induction doses), EC50 using BIS, required doses of Propofol during maintenance of anaesthesia, wake-up time.

Nature and extent of the burden and risks associated with participation benefit and group relatedness: A maximum amount of 50 milliliters of blood will be sampled from an indwelling arterial line. The patient will be asked to count slowly during induction of anaesthesia. Both induction doses of 200 and 350 milligrams are currently used standard induction doses for morbidly obese patients.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE The extreme increase of obesity in the last years had led to this study. There is no consensus about how to anaesthetise morbidly obese patients. The amounts of narcotics given during induction and maintenance of anaesthesia vary widely and rather depend on the anaesthetist than on the pharmacokinetics and dynamics in the morbidly obese patient (see figure 1 and 2). Despite the large range in induction doses (200-800 milligrams of Propofol, figure 1), the quality of induction of anaesthesia proved to be adequate in all cases. This can be explained by the central volume of distribution, which probably is the same in morbidly obese patients as in normal weight patients. This means that the induction dose of Propofol does not have to be adjusted in morbidly obese patients and that induction doses for non-obese patients can be applied, being 200 milligrams ( +/- 2.5 mg/kg). For maintenance of anaesthesia, however, pharmacokinetic parameters such as clearance and peripheral volume of distribution play an important role and are probably altered in morbidly obese patients.

   Because it is not clear how the pharmacokinetics and dynamics are affected in the morbidly obese patient, this study is performed in order to develop a population pharmacokinetic and pharmacodynamic model of Propofol when used for induction and maintenance of anaesthesia in the morbidly obese patient (BMI > 40).

   In our clinic several studies have been performed on pharmacokinetic and pharmacodynamic relations of Propofol in non-obese patients. There have been two studies on induction of anaesthesia12. One study described sedation following cardiac surgery3. There also are four studies that described sedation in the critically ill patient45 and in children67.
2. OBJECTIVES

   The study is performed in order to develop a population pharmacokinetic and pharmacodynamic model of Propofol in morbidly obese patients. A covariate analysis will be performed in order to account for variability in pharmacokinetic and pharmacodynamic parameters. The results will be used to develop individualised dosing schemes for Propofol in morbidly obese patients. This model will take into account patient and procedure bound covariates.

   Primary Objective: The main objective is to develop a pharmacokinetic model of Propofol when used for induction and maintenance of anaesthesia in the morbidly obese patient. Pharmacokinetic parameters are clearance, intercompartmental clearance, volume of central compartment and volume of peripheral compartment.

   Secondary Objective(s): The secondary objective is to develop a pharmacodynamic model of Propofol in morbidly obese patients, using the Bispectral Index and haemodynamics (heart rate and blood pressure) as a pharmacodynamic endpoint. Pharmacodynamic parameters; time to induction of anaesthesia (stop counting, eyelash reflex, quality of anaesthesia, corresponding dose required for induction of anaesthesia for both induction doses), EC50 using BIS, required doses of Propofol during maintenance of anaesthesia, wake-up time.

   A covariate analysis will be performed in order to account for variability in pharmacokinetic and pharmacodynamic parameters. Covariates: body weight, body mass index, lean body mass, length, age, PEEP and open or laparoscopic procedure, renal and hepatic function tests, haemodynamic parameters, use of co-medication.
3. STUDY DESIGN This is a randomised, therapeutic and noninvasive study, which means the whole procedure will be standard except for additional blood sampling from an indwelling arterial line during and following anaesthesia. The induction doses (200 mg or 350 mg) are both considered standard doses, as in our own survey these induction doses were found to vary between 200 and 800 milligrams (unpublished data).

Morbidly obese patients, 18-60 year old, with a Body Mass Index > 40 undergoing laparoscopic banding or gastric bypass surgery are included.

Before induction the investigators install an antecubital infusion line, an indwelling arterial blood pressure line, a Bisprectal Index (BIS) and a 3-lead ECG. The investigators give 2 millilitres of Lidocaine prior to infusion of Propofol 2 % to avoid pain during injection. Anaesthesia will be induced with a bolus of 200 milligrams or 350 milligrams of Propofol 2 % over 60 seconds delivered by a Graseby Medical 3400 pump. Patients are not given any premedication. During the bolus injection patients are asked to count. At the moment the patient stops counting a blinded observer notes the time and BIS and evaluates presence of the eyelash reflex. When the total amount of Propofol 2 % is given a blinded observer notes the BIS and presence of eyelash reflex and 250 micrograms of Fentanyl and 50 milligrams of Atracurium is given. The BIS is noted again and the patient will be intubated and mechanically ventilated. The ventilation modes are noted, as well as the amount of PEEP and when a pneumoperitoneum is used the investigators note the intra-abdominal pressure. The BIS monitors depth of anaesthesia continuously and data will be recorded at intervals of 30 seconds.

Anaesthesia is maintained by aiming at a Bispectral Index between 40 and 60. The investigators start with Propofol 2 % at an infusion rate of 25 % of total body weight (5 mg/kg/hr), with the ability to change when the aimed BIS is not reached. Remifentanyl (2 mg Remifentanyl in 40 ml of NaCl 0.9 %) and Atracurium (150 mg of Atracurium in 50 ml of NaCl 0.9 %) are standardised at infusion rates of 25 % of ideal body weight and 10 % of total body weight respectively.

Blood samples are taken from the indwelling arterial line, the exact time being recorded for each sample. At the point of sampling the investigators note the BIS. If the infusion of Propofol 2 % is changed, the time and the BIS will be noted. Extra blood samples are taken at the moment of changing the infusion rate and 5 or 15 minutes after the change in infusion rate. All samples are collected in glass oxalate tubes and analysed within three months.

At the end of the operation Propofol 2 %, Remifentanyl and Atracurium are stopped and 10 milligrams of Morphine will be given intravenously. Atracurium is antagonised with Neostigmine 1.5 milligrams and Atropine 0.5 milligrams. Postoperative pain relief is standardised with intravenous Diclofenac 3 times 75 milligrams, intravenous Paracetamol 4 times 1000 milligrams and subcutaneous Morfine 4 times 10 milligrams.

4.1 Population (base) Morbidly obese patients with a Body Mass Index > 40 undergoing laparoscopic banding or gastric bypass surgery, 18-60 year old

4.2 Inclusion criteria Patients with a Body Mass Index > 40 undergoing laparoscopic banding or gastric bypass surgery.

4.3 Exclusion criteria Epilepsy, pregnancy, breastfeeding and known allergy for Propofol, egg lecithin or soy bean oil.

4.4 Sample size calculation In this study, 20 morbidly obese patients are included. For the determination of pharmacokinetic parameters, normally 8-10 patients are required under optimal circumstances. Because the clinical situation in the operation room is less optimal compared to phase I studies in human volunteers resulting in additional variability, it is generally accepted to include 20 patients which has resulted in reliable models in previous studies from our group

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Body Mass Index > 40 undergoing laparoscopic banding or gastric bypass surgery.

Exclusion Criteria:

* Epilepsy, pregnancy, breastfeeding and known allergy for Propofol, egg lecithin or soy bean oil.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-09; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simone van Kralingen, resident, Principal Investigator — St. Antonius Hospital
Locations (1):
- st. Antonius hospital, Nieuwegein, Netherlands

REFERENCES:
- [Derived] van Kralingen S, Diepstraten J, Peeters MY, Deneer VH, van Ramshorst B, Wiezer RJ, van Dongen EP, Danhof M, Knibbe CA. Population pharmacokinetics and pharmacodynamics of propofol in morbidly obese patients. Clin Pharmacokinet. 2011 Nov 1;50(11):739-50. doi: 10.2165/11592890-000000000-00000. PMID 21973271